CLINICAL TRIAL: NCT06812832
Title: Simethicone as Part of an Enhanced Recovery After Surgery (ERAS) Protocol
Brief Title: Simethicone as Part of ERAS in Bariatric Surgery Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 971532
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-01

CONDITIONS: Simethicone; Bariatric Surgery; Post-operative Pain
Keywords: Simethicone; Gas-X; Foregut; Post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Simethicone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Arm (Placebo Comparator): This arm will receive the placebo pill
  Interventions: Drug: Placebo
- Experimental Arm (Experimental): This arm will receive simethicone
  Interventions: Drug: Simethicone 80 MG

INTERVENTIONS:
Drug: Simethicone 80 MG — Patients will receive simethicone 80mg four times per day for 2 weeks post-operatively.
  Arms: Experimental Arm
Drug: Placebo — Patients in the control group will receive a placebo pill four times per day for 2 weeks
  Arms: Control Arm

SUMMARY:
By conducting this study, we hope to assess if simethicone (also known as Gas Relief or GasX) has an effect on improving gas pain and bloating specifically in patients undergoing foregut procedures to include bariatric procedures (sleeve gastrectomy, Roux-en-Y gastric bypass), hiatal hernia, and gastric surgery.

The purpose of this research is to gather information on the safety and effectiveness of simethicone. Simethicone (more commonly known as Gas Relief or Gas-X) relieves pressure, bloating, and fullness commonly referred to as gas. It is FDA approved. The use of this medication in this research study is consistent with labeling indications.

DETAILED DESCRIPTION:
Patient enrollment Prospective participants will be screened prior to their preoperative appointment based on their presenting complaint (diagnosis) and the indicated surgical procedure (foregut operations).

Patients will undergo informed consent by a member of the research team. Patients will complete baseline survey (PROMIS Scale v1.1 - Gastrointestinal Gas and Bloating 13). This is a paper survey that will be provided to them by a member of the research team.

Patient randomization Patients will be randomized into simethicone vs placebo groups via unrestricted randomization The research pharmacist and DCI statistician will be the only individuals who know if a patient is in the experimental (simethicone) group or the control (placebo) group.

Patients will undergo their surgical procedure Postoperatively, all patients will be ordered to receive either simethicone at 80mg or placebo prepared by research pharmacist based on randomziation scheme four times per day. The research pharmacist will have the appropriate patient randomization via MRN or FIN and will provide either simethicone or placebo.

24 hours postoperatively, patients will recomplete the PROMIS Scale v1.1 - Gastrointestinal Gas and Bloating 13a for comparison as well as complete the APS Patient Outcome Questionnaire (APS-POQ-R) survey. Both of these are paper surveys that will be provided to them.

If patients are admitted for greater than 1 night, they will complete the surveys every 24 hours until discharge. These are paper surveys that will be provided to them.

Patients will be discharged with simethicone for a total of a 14 day course (to include their inpatient doses, 56 doses total) until their follow up appointment. Patients assigned to the placebo group will receive placebo (56 doses). The total number of doses any patient will receive, regardless of the length of their inpatient stay, is 56 doses. This is the number of doses total for a 14 day course when taking the medication four times per day.

At their standard postoperatively follow up visit, patients will re-complete their (PROMIS Scale v1.1 - Gastrointestinal Gas and Bloating 13a). They will also complete a compliance survey. These are both paper surveys that will be provided to them.

Data will be collected into master data sheet and data will then be de-identified with pseudo-ID assigned according to the Master Key spreadsheet. The randomization spreadsheet will only be accessed by the research pharmacist and the DCI statistician.

The master key will be kept under CAC-enabled protection The de-identified data will then be collated and analyzed Data will then be reported and submitted for relevant conferences The entirety of this project will take 4 years following IRB approval, 3 years for enrollment, perhaps an additional 1 year of data collection/analysis.

ELIGIBILITY:
Inclusion Criteria:

* Foregut procedures

Exclusion Criteria:

* Non-foregut procedures
* Allergy to simethicone
* Pregnancy or breastfeeding
* Minors under 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Pain | From enrollment through two weeks postoperatively
  Postoperative pain score - based on patient completion of the APS Patient Outcome Questionnaire (APS-POQ-R). Scores are (1) pain severity and relief; (2) impact of pain on activity, sleep, and negative emotions; (3) side effects of treatment; (4) helpfulness of information about pain treatment; (5) ability to participate in pain treatment decisions; and (6) use of nonpharmacological strategies. 0 is no pain and 10 is severe/worst pain possible. Low scores are better outcomes.
Opioid Use | Immediate post-operatively (in PACU) through 2 weeks postoperatively
  Opioid use - measured via oral morphine equivalents based on chart review and post-operative survey with patient stated opioid use after discharge
Gas and Bloating Score | From enrollment to 14 days post-operatively
  PROMIS Scale v1.0 - Gastrointestinal Reflux 13a. The PROMIS Gastrointestinal Gas and Bloating Scale includes 13 items that assess the frequency, intensity, and severity of various gastrointestinal symptoms. More specifically, the items address bloating(i.e., feeling pressure or fullness), bloating appearance (i.e., belly swollen or larger than usual size), flatulence (i.e., passing gas), and abdominal sounds (i.e., gurgling or rumbling), as well as the predictability, bothersomeness, and interference with daily activities that result from these symptoms. This measure is not disease-specific and is intended for adult respondents (ages 18+). Scores are 1-5, with 1 being "Never" and 5 being "Very Much." Low scores are better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No